CLINICAL TRIAL: NCT07241156
Title: Determining the Impact of Creative Drama on Gender Role Stress, Attitudes Toward Violence Against Women, and Aggression Among Men Affected by an Earthquake:A Randomized Controlled Trial
Brief Title: Creative Drama on Gender Role Stress, Attitudes Toward Violence Against Women, and Aggression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aslı SİS ÇELİK, Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: aslı44
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Gender Role; Aggression; Violence
Keywords: Creative Drama; Gender Role Stress; Attitudes Toward Violence Against Women; Earthquake Survivors; Men's Mental Health; Post-Disaster Psychosocial Support; Türkiye Earthquake 2023; Non-Pharmacological Intervention
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants in both the experimental and placebo groups will not be informed about which intervention they are receiving. They will be told that they are participating in different program formats as part of the same research study. The control group will receive no intervention. The data analyst/statistician, who is independent of the research team, will be blinded to group assignments. All groups (experimental, placebo, and control) will be coded as X, Y, and Z during data entry and analysis. Therefore, this study will be conducted as a double-blind design, with masking applied to the participants and the outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Experimental Group (Experimental): Participants in this group will attend 10 weekly sessions of a Creative Drama program designed to reduce gender role stress, negative attitudes toward violence against women, and aggression.
  Interventions: Behavioral: Creative Drama Program
- Arm 2 - Placebo Group (Placebo Comparator): Participants will watch 10 Turkish films over 10 weeks (one per week) containing themes of masculinity, violence against women, and aggression.
  Interventions: Behavioral: Film Viewing Sessions
- Arm 3 - Control Group (No Intervention): Participants in this group will not receive any intervention during the study period.

INTERVENTIONS:
Behavioral: Creative Drama Program — A structured 10-week Creative Drama program designed to reduce gender role stress, negative attitudes toward violence against women, and aggressive behaviors. Each session will include warm-up activities, improvisation, role-playing, and reflection components. Sessions will be conducted once a week for 90 minutes by a certified drama educator.
  Arms: Arm 1: Experimental Group
Behavioral: Film Viewing Sessions — Participants in the placebo group will watch 10 Turkish films over a 10-week period (one per week) that include themes of masculinity, gender roles, and violence. This intervention is designed as an attention-control condition to match the structure of the experimental group without providing therapeutic content.
  Arms: Arm 2 - Placebo Group

SUMMARY:
This study aims to examine the effect of Creative Drama on gender role stress, attitudes toward violence against women, and aggression among men who experienced the February 6, 2023 earthquake in Türkiye (centered in Kahramanmaraş).

A total of 75 men (25 experimental, 25 placebo, and 25 control) will participate in the study. The experimental group will take part in a creative drama program, the placebo group will watch films focusing on masculinity roles and violence for 10 weeks, and no intervention will be applied to the control group.

Data will be collected using the Gender Role Stress Scale for Men, the Attitudes Toward Violence Against Women Scale, and the Buss-Perry Aggression Questionnaire - Short Form, and will be analyzed by an independent statistician.

The study aims to enhance the psychological well-being of men affected by the earthquake in Türkiye, reduce violence against women, and contribute to gender equality.

DETAILED DESCRIPTION:
According to official reports, two major earthquakes with magnitudes of 7.7 and 7.6 occurred in Türkiye on February 6, 2023, affecting 11 provinces. The provinces of Kahramanmaraş, Hatay, Adıyaman, and Malatya were among the most severely impacted areas.

This study will be conducted as a randomized controlled experimental research to determine the effect of Creative Drama on gender role stress, attitudes toward violence against women, and aggressive behaviors among men who experienced the earthquake. The research will take place in Malatya between November 2025 and December 2026.

The study population will consist of men who experienced the Kahramanmaraş-centered earthquake on February 6, 2023, and are still residing in Malatya. The sample will include participants reached through social media platforms who meet the inclusion criteria. The data will be collected using the Participant Information Form, the Gender Role Stress Scale for Men, the Attitudes Toward Violence Against Women Scale, and the Buss-Perry Aggression Questionnaire - Short Form.

A G*Power analysis was performed to determine the sample size. Assuming a large effect size (0.80), a significance level of 0.05, and a power of 90%, it was calculated that each group should include 22 participants. Considering potential dropouts or exclusions, three additional participants per group will be added, resulting in a total of 75 participants (25 in the experimental group, 25 in the placebo group, and 25 in the control group).

Inclusion Criteria

Participants must:

Be male and volunteer to participate in the study,

Have been in Malatya during the earthquake and still reside there,

Be married during and after the earthquake,

Have no hearing or visual impairment,

Have no intellectual disability,

Have at least a primary school education,

Have no psychiatric diagnosis,

Not have received creative drama training,

Not have received psychosocial support after the earthquake,

Not have participated in any study using creative drama related to gender role stress, violence against women, or aggression,

Confirm their willingness to attend weekly sessions and comply with the program schedule.

Exclusion Criteria

Participants will be excluded if they:

Voluntarily withdraw from the study,

Fail to attend sessions regularly,

Move to another city during the study period,

Divorce during the study,

Begin receiving psychosocial support during the study period.

Randomization

The names and contact details of eligible participants will be listed. The simple randomization method will be used to ensure equal group sizes. Using the website https://www.randomizer.org/

, random numbers from 1 to 75 will be generated and divided into three groups. Three folded papers labeled with the group names will be prepared, and an independent person will randomly draw them. According to the draw, each set of 25 participants will be assigned to the corresponding group - experimental, placebo, or control - based on their position in the randomized list.

Blinding

Due to the nature of the intervention, neither the researcher nor the participants will be blinded. After completion of the study, the data from the experimental, placebo, and control groups (coded as X, Y, and Z) will be entered into a database and analyzed by an independent statistician. Therefore, the study will be conducted as a single-blind design.

Groups and Interventions

Experimental Group:

Participants will attend 10 sessions of Creative Drama, held once per week.

Placebo Group:

Participants will watch 10 Turkish films over 10 weeks (one per week) featuring themes related to masculinity roles, attitudes toward violence against women, and aggression.

Control Group:

No intervention will be applied to the participants in the control group after randomization.

ELIGIBILITY:
Inclusion Criteria:

Male individuals who experienced the 2023 Türkiye earthquake (centered in Kahramanmaraş) and currently live in Malatya.

Married during the earthquake and currently married.

Volunteer to participate in the study.

Aged between 18 and 65 years.

No hearing or visual impairments.

No intellectual disability.

At least primary school graduate.

No diagnosed psychiatric disorder.

Have not received creative drama training.

Have not received psychosocial support after the earthquake.

Have not participated in previous studies involving creative drama related to gender role stress, attitudes toward violence against women, or aggression.

Agree to attend weekly sessions and comply with the study program.

Exclusion Criteria:

Voluntary withdrawal from the study.

Failure to attend sessions regularly.

Changing residence to another city during the study period.

Divorce during the study period.

Beginning to receive psychosocial support during the study period.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only self-identified men who are biologically male, were present in Malatya during the 2023 Türkiye earthquake, and continue to live there are eligible to participate.
Enrollment: 75 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Male Gender Role Stress Levels | Baseline (Week 0) and 10 weeks after intervention
  To evaluate the effect of the Creative Drama Program on gender role stress among men who experienced the 2023 Türkiye earthquake. The Gender Role Stress Scale for Men will be used to measure changes in perceived gender-related stress.
Change in Attitudes Toward Violence Against Women | Baseline (Week 0) and 10 weeks after intervention
  To assess the impact of the Creative Drama Program on men's attitudes toward violence against women. The Attitudes Toward Violence Against Women Scale will be administered to measure changes in participants' beliefs and attitudes.
Change in Aggression Levels | Baseline (Week 0) and 10 weeks after intervention
  To determine the effect of the Creative Drama Program on aggression among male earthquake survivors. The Buss-Perry Aggression Questionnaire - Short Form will be used to assess total aggression and subscale scores (physical aggression, verbal aggression, anger, and hostility).

CONTACTS AND LOCATIONS:
Overall Officials: Aslı SİS ÇELİK, Study Director — Ataturk University

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to ethical considerations and the sensitivity of personal information collected from earthquake survivors. Only aggregated results will be published in scientific journals.

DOCUMENTS (1):
  • Study Protocol (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT07241156/Prot_000.pdf